CLINICAL TRIAL: NCT04630717
Title: Effect of an Hypnotherapy Right Before the Induction of Anesthesia Versus Standard Induction on NOL Variations After Standardized Stimulation Performed Under General Anesthesia The HYPNOSTIMNOL Study
Brief Title: Effect of an Hypnotherapy Session on the NOL Variations After Stimulation
Acronym: HYPNOSTIMNOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, MD, PhD, Professor, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-2446
Record Dates: First submitted 2020-10-28; First posted 2020-11-16 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Anesthesia; Hypnosis; Pain
Keywords: Hypnosis; Anesthesia; Pain; Nociception; NOL
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Prospective randomized double-blind, single-center trial. The patient does not know whether or not he is in the "hypnotic conversation" group; nor does the anesthesiologist managing the patient intraoperatively knows whether or not the patient had a hypnotic conversation prior to general anesthesia induction.
Who Masked: Participant, Care Provider
Masking Description: Prospective randomized double-blind, single-center trial. The patient does not know whether or not he is in the "hypnotic conversation" group; nor does the anesthesiologist managing the patient intraoperatively knows whether or not the patient had a hypnotic conversation prior to general anesthesia induction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): normal discussion before general anesthesia induction
  Interventions: Other: control groupe
- Hypnosis group (Active Comparator): hypnosis session before general anesthesia induction
  Interventions: Other: Medical hypnosis session

INTERVENTIONS:
Other: Medical hypnosis session — the therapist will use a standard and identical protocol in all patients: the International characteristics of the hypnosis protocol are the following hypnotic induction through conversational hypnosis and interviewing about leisure activity.
  A catalepsy of the hand or the finger will be done, also to stabilize hypnosis if it is accepted by the patient
  Arms: Hypnosis group
Other: control groupe — the therapist will use usual voice,loud and strong voice,. clear, high position of the doctor, medical speech focused,no question about the patient's privacy will be made.
  Arms: control group

SUMMARY:
The investigators propose to evaluate the analgesic effect of medical hypnosis prior to the pharmacological induction of general anesthesia versus a classical pharmacological induction of anesthesia. Monitoring of the NOL index (Nociception index) as well as all the other classical parameters under general anesthesia (heart rate, blood pressure etc) will allow evaluation of the level of nociception related to oro-tracheal intubation as well as the one related to standardized electrical tetanic stimulation during general anesthesia and before surgical incision, between the two groups.

The investigators know from the literature that the use of medical hypnosis in combination with anesthetic drugs allows for a significant reduction of hypnotic and opioid drugs.

The investigators aim here at evaluating the real and objective impact of pre-anesthesia hypnosis on intraoperative nociception by using the NOL index which has been developed and used recently to better detect nociceptive stimuli under anesthesia.

This clinical trial will provide an objective answer on the analgesic properties of intraoperative hypnosis. If this is confirmed, hypnosis could find its place in the management of perioperative nociception around general anesthesia.

DETAILED DESCRIPTION:
Study Design: Prospective randomized double-blind, mono-centric trial (patient does not know if the conversation is hypnotic or not, the anesthesiologist in charge during the case is not here during the preoperative conversation and is not the one doing the medical conversational hypnosis or standard conversation).

This study proposes to answer two questions :

* To measure the difference in the variation of the NOL index (delta NOL) after standardized electrical stimulation performed after tracheal intubation under general anesthesia between two types of anesthetic induction : pharmacological induction associated with a brief session of medical hypnosis versus a standard pharmacological induction.
* To measure variation of heart rate, arterial pressure, BISpectral index after intubation, standardized electrical stimulation, incision and other intraoperative surgical stimuli. Evaluation of postoperative pain, analgesic consumption in the recovery room, and recovery room discharge time.

  50 Adults scheduled for elective laparoscopic surgery under general anesthesia expected to last less than 3 hours will be enrolled.

Patients will be informed and included the day before surgery. Randomization will be done by web-base-systeme-algorithm dividing patients into two groups: general anesthesia alone or general anesthesia coupled with hypnosis. No premedication will be administered.

The hypnotherapist will meet briefly with the patient before admission to the operating room to introduce himself.

When the patient enters the operating room, a checklist is performed by the staff, the usual monitoring is set up (electrocardiogram, pulse oximeter, non-invasive blood pressure, muscle relaxation monitor, bispectral index, NOL index). Nasoparyngeal temperature and monitoring of expired carbon dioxide will be placed following tracheal intubation to allow monitoring of normothermia and normo capnia intraoperatively.

The PMD200TM monitor and the BIS index will be connected to the patient. Registration of the index NOL will be done continuously via the PMD200TM monitor, which will be switched on at the start of the procedures.

When everything is ready for pharmacological induction the anesthesiologist in charge will leave the operating room.

In the control arm the therapist will have a standard discussion to check all things are all right with the patient before pharmacological induction starts. No hypnotic conversation will be proposed.

In the hypnosis arm a short session of hypnosis will be done before the pharmacological induction.

The period of discussion in both the groups will be between 6 and 15 minutes, hypnotic or not.

Then, the anesthesiologist will be called for pharmacological induction of general anesthesia.

The protocol of anesthesia will be the same in both groups : the induction will be done by propofol (with a goal of Bispectral index : 40-60) and Remifentanil (with goal of NOL < 25), and muscle relaxation with Rocuronium (0.8 mg.kg-1).

After tracheal intubation, the remifentanil will be discontinued. After a period of at least 10 minutes after remifentanil discontinuation, a standardized tetanic stimulation (70mA, 100Hz, 30 seconds at the ulnar level) will be applied and all the anesthesia parameters and NOL index will be electronically recorded every 5 seconds.

After this stimulation, general anesthesia will be maintained as follows: sevoflurane inhaled anesthesia for a bispectral index between 40-60; remifentanil analgesia for a NOL index between 5-25; rocuronium for a muscle relaxation with TOF index between 1-3. Total consumption of remifentanil during the case will be monitored and calculated in mcg.kg-1 per hour of surgery as it will be a surrogate of intraoperative pain/nociception that will be analyzed too. At the end of surgery, anesthesia is discontinued, hydromorphone 7mcg.kg-1 will be administered at the end of skin closure in anticipation of postoperative pain. Acetaminophen will also be given PR at the end of surgery as well as intravenous ketorolac. Skin incisions for laparoscopic surgery will be infiltrated with 0.5% bupivacaine (maximum 20mL). Once the patient extubated, she/he will be transferred to post anesthesia care unit (PACU) where classical pain management will be offered. Pain scores in PACU, patients' satisfaction, opioid consumption will be evaluated between the two groups in PACU.

Data analysis: The main outcome analyzed will be the delta NOL or the variation of the NOL index between pre and post stimulation in the two groups. The mean maximum value of the NOL index after stimulation will also be compared between the two groups.

Statistical analyses will be performed using SAS version 9.4 or higher and will be performed at a bilateral significance level of 0.05, unless otherwise specified. Descriptive statistics of central tendency (e.g., mean and 95% CI, median) and dispersion (SD, frequency table) will be used to describe the characteristics of the patients in each group of the study. The intraoperative data collected in the groups will be compared using parametric (e.g. Student's t-test) or non-parametric (e.g. Mann-Withney's U-test, Chi-square test) tests depending on the type of variables and their distribution.

ELIGIBILITY:
Inclusion Criteria:

* ASA score I, II or III
* Age 18 years or older
* Elective laparoscopic surgery under general anesthesia duration less than 3 hours
* Good understanding of French
* Acceptance of the protocol

Exclusion Criteria:

* Emergency Surgery
* Pregnant or breastfeeding woman
* Pre-operative hemodynamic failure
* Pathologies of the central nervous system (traumatic sequelae, epilepsy, mental retardation)
* Dependence on drugs or alcohol in the last 6 months
* Consumption of chronic psychotropic drugs for more than 3 months
* Morphine consumption or chronic pain requiring a morphine equivalent of 20 mg po daily for more than 6 weeks.
* Psychiatric pathologies
* Patient Refusal
* Allergy or intolerance to one of the products in the study

Exclusion criteria :

* Difficult planned and unplanned intubation
* Unexpected intraoperative complications (circulatory failure, hemorrhage, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Delta NOL (no unit for the NOL index) | From 1 minute before to 3 minutes after the tetanic stimulation for each patient under general anesthesia
  To compare the variation of NOL (delta NOL) after tetanic stimulation under general anesthesia based on hypnosis versus standard care group

SECONDARY OUTCOMES:
Delta Heart Rate (beat per minute) | From 1 minute before to 3 minutes after the tetanic stimulation for each patient under general anesthesia
  To compare the variation of heart rate (HR) after tetanic stimulation under general anesthesia based on hypnosis versus standard care group
Delta Mean Arterial Blood Pressure (unit:mmHg) | From 1 minute before to 3 minutes after the tetanic stimulation for each patient under general anesthesia
  To compare the variation of mean arterial blood pressure (MABP) after tetanic stimulation under general anesthesia based on hypnosis versus standard care group
Delta BIS (no unit for BIS index) | From 1 minute before to 3 minutes after the tetanic stimulation for each patient under general anesthesia
  To compare the variation of bispectral index (BIS) after tetanic stimulation under general anesthesia based on hypnosis versus standard care group
Peak value of NOL (no unit) | From 1 minute before to 3 minutes after the tetanic stimulation for each patient under general anesthesia
  To compare the peak value of NOL after tetanic stimulation under general anesthesia based on hypnosis versus standard care group
Area Under the Curve (AUC) for NOL (no unit) | From T0 (start stimulation) to 3 minutes after tetanic stimulation for each patient
  To compare the AUC of NOL after tetanic stimulation under general anesthesia based on hypnosis versus standard care group
Total Dose of Remifentanil (unit: mcg) | Intraoperative]
  Total dose of remifentanil in mcg from induction of anesthesia until tracheal extubation
Total Dose of Hydromorphone in post-anesthesia care unit (PACU) (unit: mg) | From entrance in PACU until discharge, an average of 2 hours
  Total dose of hydromorphone (mg) in PACU
Pain Scores (scale from 0 to 10) in PACU | From entrance in PACU until discharge, an average of 2 hours
  Maximum Pain scores in PACU
Postoperative nausea and vomiting (PONV) score (scale from 0 to 3) in PACU | From entrance in PACU until discharge, an average of 2 hours
  PONV score on a scale from 0 (none nausea and vomiting ) to 3 (maximum nausea and vomiting ) in PACU
Pasero Opioid-Induced Sedation Scale (POSS score) (scale from 1 to 4) in PACU | From entrance in PACU until discharge, an average of 2 hours
  POSS score on a scale from 1 (sleep, easy to arouse ) to 4 (somnolent, minimal or no response) in PACU
Time for PACU discharge based on Aldrete score (scale from 0 to 10) (in minutes) | From entrance in PACU until discharge, an average of 2 hours
  Time (in minutes) for readiness for PACU discharge based on Aldrete score greater than or equal to 9

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No